CLINICAL TRIAL: NCT03212703
Title: A Trial of Mindfulness-Based Skills Training Groups Versus a Waiting List Control Period for Parents of Obsessive-Compulsive Disorder (OCD)-Affected Youth
Brief Title: Mindfulness for Parents of OCD-affected Children
Acronym: MBST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Evelyn Stewart, MD, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-02099
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Mindfulness training; Parents and families; Pediatric OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (WLC) (Active Comparator): Observation surveys over an 8-week period.
  Interventions: Behavioral: Mindfulness-Based Skills Training (MBST)
- Mindfulness-Based Skills Training (MBST) (Active Comparator): Attendance at weekly 1.5-hour group sessions and surveys over an 8-week period.
  Interventions: Other: Waitlist control (WLC)

INTERVENTIONS:
Behavioral: Mindfulness-Based Skills Training (MBST) — 8-week mindfulness skills training sessions based on Mindfulness-Based Cognitive Therapy (MBCT) program by Zindel Segal, Mark Williams and John Teasdale
  Arms: Waitlist control (WLC)
Other: Waitlist control (WLC) — Observation surveys at baseline, mid-point and end-point of an 8-week period
  Arms: Mindfulness-Based Skills Training (MBST)

SUMMARY:
The purpose of this study is to investigate the role of a mindfulness-based skills training program for parents of children with obsessive compulsive disorder (OCD). The investigators will explore if parents involved in this group experience any change in their levels of stress, feelings of being an effective parent and family relationships compared to a waiting list control period. The investigators will look at how the family manages OCD in their lives. In particular, if mindfulness skills training will help increase the parents ability to tolerate distress in their child secondary to OCD and as such reduce the family accommodation of OCD. As family accommodation is an important negative prognostic predictor for children with OCD, changes in OCD symptom severity and functional impact in these child will also be measured.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a debilitating psychiatric illness that frequently begins in childhood. It is characterized by obsessions and/or compulsions that are distressing, time consuming and significantly impairing. OCD is distinct in the extent to which it disrupts family functioning, in that there is intense parental pressure to become involved in rituals and to change home environments and schedules to avoid triggers, thus accommodating the OCD. It is also well known that OCD severity tends to worsen in the context of stressful environments and situations. While effective treatment approaches for pediatric OCD have been identified, partial response and treatment refusal are all too common, leading to chronicity of both the illness itself and of its deleterious familial effects.

The investigators plan to study a novel approach to help manage the stress of parenting a child with OCD, thus facilitating more effective resistance to OCD family accommodation and supporting the child in fighting this difficult illness. The investigators will explore the role of group-based mindfulness-based skills training (P-MBST) in supporting parents of OCD-affected youth, in particular investigating the possibility that increased distress tolerance as a result of mindfulness practice may help parents reduce OCD accommodation.

ELIGIBILITY:
Inclusion Criteria:

1. Parents (or step-parents or legal guardians) with care-giving role for an OCD-affected youth from our clinic
2. Participants must be able to converse in English
3. Participants willing to attend 8 sessions of a weekly 1.5 hour group, in addition to complete questionnaires at multiple time points during the group and waiting list period.

Exclusion Criteria:

1. Parents who have previously participated in mindfulness skills training.
2. Parents with active psychosis, mania, mental retardation, autism or current substance misuse.
3. Parents unwilling to provide consent.
4. Families who are not attending our program's group-family Cognitive-Behavioral Therapy treatment concurrently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change in parental stress levels compared to waiting list control (WLC). | Baseline (first week of P-MBST), Mid-treatment (fifth week of P-MBST), Post-treatment (within one week of completing 8-week P-MBST sessions) and follow-up (one month following P-MBST)
  Parental stress levels is measured using the Parenting Stress Index - Short Form (PSI-SF) for parents with children under 13 years of age and the Stress Index for Parents of Adolescents - Short Form (SIPA-SF) for parents with children who are 13 years and older. The PSI-SF and SIPA-SF are both measures of parental stress, but with a difference in age cut-off.
Change in ability to tolerate OCD-related distress compared to waiting list control (WLC). | Baseline (first week of P-MBST), Mid-treatment (fifth week of P-MBST), Post-treatment (within one week of completing 8-week P-MBST sessions) and follow-up (one month following P-MBST)
  The ability to tolerate OCD-related distress is measured using the Parental Tolerance of Child Distress (PT-OCD) scale.

SECONDARY OUTCOMES:
Change in ability to resist family accommodation of the child's OCD symptoms compared to waiting list control (WLC). | Baseline (first week of P-MBST), and Post-treatment (within one week of completing 8-week P-MBST sessions).
  Family accommodation is measured by the Family Accommodation Scale (FAS)
Change in family functioning compared to the waiting list control (WLC). | Baseline (first week of P-MBST), and Post-treatment (within one week of completing 8-week P-MBST sessions).
  Family functioning in relation to the impact of OCD on the family is measured by the OCD Family Functioning Scale (OFF).
Change in OCD severity compared to waiting list control (WLC). | Baseline (first week of P-MBST), and Post-treatment (within one week of completing 8-week P-MBST sessions).
  OCD symptom severity is measured with the Children's Yale Brown Obsessive-Compulsive Scale (CY-BOCS), rated by the parent.
Change in OCD-associated coercive and disruptive symptoms compared to waiting list control (WLC). | Baseline (first week of P-MBST), and Post-treatment (within one week of completing 8-week P-MBST sessions).
  Coercive and disruptive behaviours is measured using the Coercive and Disruptive behaviours in Pediatric OCD (CD-POC) scale.

OTHER OUTCOMES:
Change in mindfulness compared to waiting list control (WLC). | Baseline (first week of P-MBST), and Post-treatment (within one week of completing 8-week P-MBST sessions).
  The Mindfulness Personality Profile (MPP) will be used to assess Mindfulness over the following four domains:
  1. Self-description - adapted from the Self-Description Questionnaire (Marsh, 1994)
  2. Awareness and attention - adapted from Mindfulness Attention Awareness Scale (Brown and Ryan, 2003)
  3. Self-compassion and time - adapted from the Self-Compassion Scale (Raes et al., 2011) and Adolescent Time Inventory (Mellow and Worrell, 2007; Mello et al., 2013)
  4. Self reflection and insight scale (SRIS) ((Grant, Fraknlin and Langford, 2002)

CONTACTS AND LOCATIONS:
Overall Officials: S. Evelyn Stewart, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Belschner L, Lin SY, Yamin DF, Best JR, Edalati K, McDermid J, Stewart SE. Mindfulness-based skills training group for parents of obsessive-compulsive disorder-affected children: A caregiver-focused intervention. Complement Ther Clin Pract. 2020 May;39:101098. doi: 10.1016/j.ctcp.2020.101098. Epub 2020 Jan 17. PMID 32379640